CLINICAL TRIAL: NCT04812769
Title: Electronic Consultation for AD/ADRD Residents Experiencing Infectious Diseases
Acronym: eCARE-ID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is taking a leave of absence. Study terminated.
Sponsor: Yale University (Other)
Collaborators: Advarra (Industry); National Institute on Aging (NIA) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000029812; RFA-IMPACT-20-P02A (Other Grant/Funding Number: NIA); U54AG063546 (NIH)
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer's Dementia; Nursing Homes; Antibiotics; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two participating nursing homes will be assigned to the intervention. One participating nursing home will serve as a control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Two nursing homes will receive the eCARE-ID intervention
  Interventions: Device: eCARE-ID
- Control (Placebo Comparator): One control nursing home will receive infectious disease consultations and antibiotic stewardship services per routine practice.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: eCARE-ID — The intervention, eCARE-ID, consists of: 1) telehealth video clinical consultation services for nursing homes residents; 2) electronic consultation services for healthcare personnel; 3) telehealth video antibiotic stewardship services for healthcare personnel
  Arms: Intervention
Other: Standard of Care — Standard of care will be delivered to the control home.
  Arms: Control

SUMMARY:
Pilot study to evaluate the feasibility of a pilot embedded pragmatic cluster randomized controlled trial to reduce the duration of antibiotic therapy and number of antibiotic prescriptions in nursing home residents with AD/ADRD.

DETAILED DESCRIPTION:
The overall objective of the proposed investigation is to assess the feasibility of a pilot embedded pragmatic cluster randomized controlled trial (ePCT) to reduce the duration of antibiotic therapy and number of antibiotic prescriptions among nursing home residents with AD/ADRD. With the support of three independently owned and operated nursing homes that are unaffiliated with an academic medical center, we have developed the multicomponent intervention, eCARE-ID (Electronic Consultation for AD/ADRD Residents Experiencing Infectious Diseases). eCARE-ID consists of three components: 1) Tele-ID video clinical consultation services for nursing home residents; 2) electronic consultation (e-consultation) services for healthcare personnel at participating nursing homes; and 3) Tele-ID video antibiotic stewardship services for healthcare personnel including pharmacists at participating nursing homes.

ELIGIBILITY:
Inclusion criteria - residence in a participating nursing home

Exclusion criteria:

- Not willing to consent to the study

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic therapy in nursing home residents | 6 months
  The primary outcome will be defined as the duration of antibiotic therapy in nursing home residents with AD/ADRD, measured as the total days of antibiotic therapy per 1000 resident-days among residents with ADRD.

SECONDARY OUTCOMES:
Number of antibiotic prescriptions in nursing home residents | 6 months
  The secondary outcome will be defined as the number of antibiotic prescriptions in nursing home residents with AD/ADRD, defined as the total number of antibiotic prescriptions per 1000 resident-days among residents with AD/ADRD.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Juthani-Mehta, M.D., Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No